CLINICAL TRIAL: NCT03409653
Title: Complex Chronic Diseases Program Data Registry
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: BC Women's Hospital & Health Centre (Other)
Collaborators: Ministry of Health, Province of British Columbia (Unknown)
Responsible Party: Principal Investigator, Luis Nacul, Medical Director CCDP, Complex Chronic Care Clinic, BC Women's Hospital & Health Centre
Other Study IDs: H16-01648
Record Dates: First submitted 2017-11-30; First posted 2018-01-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Fibromyalgia; Chronic Fatigue Syndrome; Myalgic Encephalomyelitis; Chronic Lyme-Like Syndrome
Keywords: fatigue; pain; chronic pain; Data registry; ME/CFS; CFS; FM; Post-exertional malaise; Lyme
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic; Fatigue; Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this data registry is to prospectively collect data from patients referred to an Complex Chronic Diseases Program (CCDP) at BC Women's Hospital + Health Centre to assess the quality of life of the CCDP Patients before, during and after their care at the CCDP.

DETAILED DESCRIPTION:
1. Before their initial intake appointment, all CCDP patients are given a patient binder that includes the baseline Standardized Questionnaires. These are clinical questionnaires that all patients complete regardless of whether or not they consent to participation in research. In addition to the questionnaires completed at baseline, patients who consent to participate in the data registry will complete the questionnaires, via email or paper copy, at the following time points: approximately 6 months after intake, at discharge and 3 months post-discharge.
2. Patients who consent to the data registry will also be asked to complete a short questionnaire collecting basic demographic information at baseline. The demographic questionnaire will be either mailed to their home or sent via an online link; the investigators will ask participants to complete this form either before or when they come in for their first in-person visit at the CCDP.
3. Additional data will be collected and entered from the clinical chart. Specifically, after the patient's initial clinic appointment, the Research Coordinator or designate will enter data points from the Interdisciplinary Assessment Tool, into REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Newly referred patients of the Complex Chronic Diseases Program
* Must be able to read and understand English
* 18 years of age or older

Exclusion Criteria:

* Have not completed the Standardized Questionnaires booklet prior to the initial intake assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Complex Chronic Diseases Program at BC Women's Hospital + Health Centre all have signs, symptoms or a diagnosis of: Fibromyalgia (FM), Chronic Fatigue Syndrome/Myalgic Encephalomyelitis (ME/CFS), and/or Chronic Lyme-Like Syndrome (CLLS).
  The factors involved in causing all three of these diseases are not well understood (Jain et al. 2003, Wolfe et al. 2010, Carruthers et al. 2003). Furthermore, symptoms, severity of symptoms and the effects of all of these complex chronic diseases can vary greatly among people with the same diagnosis.
  All of these conditions are currently diagnosed according to the particular group of symptoms described by the patient.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life | Baseline (pre-intake), 6 months, discharge (an average of 21 months), 3 months post-discharge
  Change in self-reported quality of life assessed by structured questionnaire (36 Item Short Form Health Survey (SF-36))

SECONDARY OUTCOMES:
Brief Pain Inventory Short Form (BPI-SF) | Baseline (pre-intake), 6 months, discharge (an average of 21 months), 3 months post-discharge
  The BPI-SF is a self-reported standard questionnaire used to evaluate the severity of pain and the impact of this pain on the patient's daily functioning.
Fatigue Severity Scale (FSS) | Baseline (pre-intake), 6 months, discharge (an average of 21 months), 3 months post-discharge
  The FSS is a self-reported standard questionnaire that uses a scale to measures the severity of the fatigue and its effect on a person's activities and lifestyles in patients with a variety of disorders. It uses a 7- point Liker scale, where 1=Strongly Disagree and 7= Strongly agree. Score range is 1-7. Higher schore indicates more severe fatigue.
McGill Pain Questionnaire Short Form | Baseline (pre-intake), 6 months, discharge (an average of 21 months), 3 months post-discharge
  The McGill Pain Questionnaire Short Form is self-reported standard questionnaire. It is used to describes the subjective overall intensity of the total pain experience.
Pittsburgh Sleep Quality Index (PSQI) | Baseline (pre-intake), 6 months, discharge (an average of 21 months), 3 months post-discharge
  The PSQI is a self-reported standard questionnaires. It is used to assess sleep quality and disturbances.
Patient Health Questionnaire 9 (PHQ - 9) | Baseline (pre-intake), 6 months, discharge (an average of 21 months), 3 months post-discharge
  The PHQ-9 is a self-reported standard questionnaire used to screen, diagnose, monitor and measure the severity of depression.
Generalized Anxiety Disorder - 7 item (GAD - 7) | Baseline (pre-intake), 6 months, discharge (an average of 21 months), 3 months post-discharge
  The GAD-7 is a self-reported standard questionnaire used to measures the severity of various signs of general anxiety disorder according to response categories with assigned points.

CONTACTS AND LOCATIONS:
Overall Officials: Luis C Nacul, MD, Principal Investigator — Medical Director CCDP, Complex Chronic Care Clinic; Wee-Shian Chan, MD, Study Chair — Department Head, Medicine
Locations (1):
- BC Women's Hospital + Health Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No